CLINICAL TRIAL: NCT04464447
Title: Feasibility of Group-based Acceptance and Commitment Therapy for Adolescents (AHEAD) With Functional Somatic Syndromes: A Pilot Study
Brief Title: Feasibility and Pilot Testing of Group-based ACT for Adolescents With Functional Somatic Syndromes
Acronym: AHEAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD pilot
Record Dates: First submitted 2020-06-27; First posted 2020-07-09 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2020-06

CONDITIONS: Functional Disorder
MeSH Terms: interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group-based Acceptance and Commitment Therapy (Other): Group-based Acceptance and Commitment Therapy (ACT) for adolescents presenting with multiple functional somatic syndromes.
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — The treatment "ACT for Health in Adolescents" (AHEAD) is an ACT-based Group intervention consisting of 9 modules (27 hours in total) delivered over a period of 3 months, with a follow-up meeting (3 hours) 3 months after the last module. Six to eight patients participate in each treatment Group. An information meeting (3 hours) for close relatives is held at the beginning of the Group treatment and the adolescents and their parents were invited to a 1½-hour individual consultation after the 8th module.

SUMMARY:
Recurrent and impairing functional somatic syndromes (FSS) are common in adolescents. Despite a high need for care, empirically supported treatments are lacking for youth. The aim of the uncontrolled was to assess feasibility and treatment potential of group-based Acceptance and Commitment Therapy (ACT) in a generic treatment approach for adolescents with multiple FSS i.e. "ACT for Health in Adolescents" (AHEAD).

ELIGIBILITY:
Inclusion Criteria:

* Bodily Distress Syndrome, multi-organ type of at least 12 months' duration
* Raised since early childhood in Denmark or born by Danish parents
* Understand, speak and read Danish
* Moderate or severe impairment

Exclusion Criteria:

* Acute psychiatric disorder demanding other treatment, or if the patient is suicidal.
* A lifetime diagnosis of psychosis, mania or depression with psychotic symptoms (ICD-10: F20-29, F30-31, F32.2, F33.3), serious cognitive deficits or developmental disorders such as mental retardation and autism (ICD-10: F70, F84)
* Substance abuse of e.g. narcotics, alcohol or medication.
* Pregnancy at time of inclusion
* Not able to participate in group-based treatment, e.g. patients with severe ADHD (ICD-10: F90), severe social phobia (ICD-10: F40.1) or conduct disorder (ICD-10: F91)

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2013-05-29 (Actual); Primary Completion 2015-04-15 (Actual); Study Completion 2015-04-24 (Actual)

PRIMARY OUTCOMES:
Change in Short Form Health Survey-36 (SF36) (Assessment of an aggregate score measuring physical health) | At baseline (i.e. at clinical assessment), and at 2, 4, 5, and 8 months (corresponding to group start, 8th, 9th module and follow up meeting)
  Questionnaire, patient rated. Physical health measured with aggregate scores of the scales PF (physical functioning), BP (bodily pain) and VT (vitality). Score range 15-65. Higher scores indicating a higher degree of self-rated physical health.

SECONDARY OUTCOMES:
Change in Bodily Distress Syndrome checklist (BDS checklist) | At baseline (i.e. at clinical assessment), and at 2, 4, 5, and 8 months (corresponding to group start, 8th, 9th module and follow up meeting)
  Questionnaire, patient rated. Assessment of symptom severity. Score range 0-100. Higher score indicating a higher degree of symptom severity.
Change in Limitation index Questionnaire | At baseline (i.e. at clinical assessment), before psychiatric consultation (approximately 2 weeks after clinical assessment), and at 2, 3, 4, 5, and 8 months (corresponding to before therapy, after 4th, 8th, 9th module and at follow up meeting)
  Questionnaire, patient rated. Assessment of symptom interference. Score range 0-36 with higher score indicating a higher degree of limitation.
Change in Whiteley 7 | At baseline (i.e. at clinical assessment), and at 2, 4, 5, and 8 months (corresponding to group start, 8th, 9th module and follow up meeting)
  Questionnaire, patient rated. Assessment of illness worry. Overall mean item score range from 0-4 with higher scores indicating a higher degree of illness worry.
Change in SCL-8 Questionnaire | At baseline (i.e. at clinical assessment), and at 2, 4, 5, and 8 months (corresponding to group start, 8th, 9th module and follow up meeting)
  Questionnaire, patient rated. Assessment of emotional distress. Overall mean score range from 0-4 with higher scores indicating a higher degree of emotional distress.
Change in SF-36 PCS | At baseline (i.e. at clinical assessment), and at 2, 4, 5, and 8 months (corresponding to group start, 8th, 9th module and follow up meeting)
  Aggregate score from questionnaire - physical component summary. Patient rated. The aggregate score has a mean of 50 and a SD of 10, but no range. Higher scores indicate better physical health.
Change in SF-36 MCS | At baseline (i.e. at clinical assessment), and at 2, 4, 5, and 8 months (corresponding to group start, 8th, 9th module and follow up meeting)
  Aggregate score from questionnaire - mental component summary. Patient rated. The aggregate score has a mean of 50 and a SD of 10, but no range. Higher scores indicate better mental health.
Change in IPQ-R Illness Perceptions Questionnaire | At baseline (i.e. at clinical assessment) and at 2, 3, 4, 5, and 8 months (corresponding to before therapy, after 4th, 8th, 9th module and at follow up meeting)
  Questionnaire, patient rated. Treatment target. Score range 0-80 with higher scores reflecting a more maladaptive view of the illness.
Change in BRIQ Behavioural Responses to Illness Questionnaire | At baseline (i.e. at clinical assessment) and at 2, 3, 4, 5, and 8 months (corresponding to before therapy, after 4th, 8th, 9th module and at follow up meeting)
  Questionnaire, patient rated. Assessment of illness related behaviour. Treatment target. Measures two dimensions of illness behaviour i.e. limiting behaviour (score range 7-35) and all-or-nothing behaviour (score range 6-30). Higher scores indicate a higher degree of maladaptive behaviour.
Change in AFQ-Y8 (Avoidance and Fusion Questionnaire in Youth) | At baseline (i.e. at clinical assessment) and at 2, 3, 4, 5, and 8 months (corresponding to before therapy, after 4th, 8th, 9th module and at follow up meeting)
  Questionnaire, patient rated. Assessment of psychological flexibility. Treatment target. Score range 0-32 with higher scores relfecting a higher degree of psychological inflexibility.
PGIC (Patient Global Impression of Change) | At 8 months corresponding to at follow up meeting
  Questionnaire, patient rated. 7 point scale with answers ranging from "no change or condition gotten worse" to "a great deal better and a considerable improvement that has made all the difference".

OTHER OUTCOMES:
Modified version of ESQ Experience of Service Questionnaire | At 8 months corresponding to at follow up meeting
  Questionnaire, patient rated. Assessment of their treatment experience.
Questions concerning close relatives' satisfaction with information meeting | At meeting for close relatives corresponding to approximately 1 week after start of group therapy (i.e. at 2 months)
  Questions regarding specific meeting content and possibility of free text comments. Rated by close relatives.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte U Rask, MD, PhD, Principal Investigator — Aarhus University and during study the Research Clinic for Functional Disorders and Psychosomatics

IPD SHARING:
Plan to Share IPD: No
Has not been incorporated in the consent from the patients. However, some data will be available upon request.

REFERENCES:
- [Derived] Kallesoe KH, Schroder A, Wicksell RK, Preuss T, Jensen JS, Rask CU. Feasibility of group-based acceptance and commitment therapy for adolescents (AHEAD) with multiple functional somatic syndromes: a pilot study. BMC Psychiatry. 2020 Sep 21;20(1):457. doi: 10.1186/s12888-020-02862-z. PMID 32957944